CLINICAL TRIAL: NCT03576248
Title: Effect of Transcranial Electrical Stimulation on the Consciousness of Non-communicating Patients.
Brief Title: CONsciousness Transcranial Electric STimulation
Acronym: CONTEST_3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expected number of patients unreached because of COVID19 pandemics. Inclusion stopped at N=20 patients (lower expected number of patients).
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C17-56; 2017-A02763-50 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2019-01

CONDITIONS: Disorder of Consciousness
Keywords: State of consciousness; tACS; tDCS; Global neuronal workspace; Brain injury
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This study is composed of two independent sub-studies, one exploring the effects of tACS and the other the effects of tDCS, with different participants assigned to the two sub-studies. There will be 2 arms in tACS group and 2 arms in tDCS group. Among each sub-study, all participants will participate in all arms (hence the cross-over design).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study will be double-blind : neither participant nor the investigator will know which stimulation type (in-phase active, anti-phase active or sham) is on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- In-phase 6 Hz prefronto-parietal tACS (Experimental): 6 Hz stimulation (1000 μA) with transcranial Alternative Current Stimulation (tACS) will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3 of the 10-20 international scalp EEG system, with a return electrode in Cz) for 20 minutes. The phase difference between the two stimulation sites will be 0°.
  Interventions: Device: In-phase 6 Hz prefronto-parietal tACS
- Sham prefronto-parietal tACS (Sham Comparator): The same stimulation as in in-phase transcranial Alternative Current Stimulation tACS (6 Hz F3 and P3 stimulation with 0° phase difference) will start with a current intensity of 1000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. The whole session duration is 20 minutes.
  Interventions: Device: Sham prefronto-parietal tACS
- 2 mA left prefrontal tDCS (Experimental): 2000 μA anodal transcranial Direct Current Stimulation (tDCS) will be applied over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system with a right supraorbital return electrode (Fp2 of the 10-20 international scalp EEG system) during 20 minutes.
  Interventions: Device: 2 mA left prefrontal tDCS
- Sham left prefrontal tDCS (Sham Comparator): The same stimulation as active transcranial Direct Current Stimulation (tDCS) (anodal F3 and return in Fp2) will start at 2 mA intensity for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. The whole session duration is 20 minutes.
  Interventions: Device: Sham left prefrontal tDCS

INTERVENTIONS:
Device: In-phase 6 Hz prefronto-parietal tACS — tACS is a non-invasive stimulation technique that works by delivering a weak sinusoidally oscillating electrical current to the surface of the skull to entrain oscillations in the brain.
  Arms: In-phase 6 Hz prefronto-parietal tACS
Device: Sham prefronto-parietal tACS — tACS is a non-invasive stimulation technique that works by delivering a weak sinusoidally oscillating electrical current to the surface of the skull to entrain oscillations in the brain.
  Arms: Sham prefronto-parietal tACS
Device: 2 mA left prefrontal tDCS — tDCS is a form of neuromodulation method where very low levels of constant current are delivered to specifically targeted areas of the brain
  Arms: 2 mA left prefrontal tDCS
Device: Sham left prefrontal tDCS — tDCS is a form of neuromodulation method where very low levels of constant current are delivered to specifically targeted areas of the brain
  Arms: Sham left prefrontal tDCS

SUMMARY:
The aim of this study is to investigate the effect of transcranial Alternating Current Stimulation (tACS) at theta frequency and the the effect of transcranial Direct Current Stimulation (tDCS) on the conscious state of non-communicating patients. tACS and tDCS are non-invasive stimulation techniques that are used to induce brain oscillations at certain frequency or to increase the brain activity in applied region.

Limited treatments are available to improve consciousness in severely brain injured patients. Transcranial Direct Current stimulation (tDCS) is one of the few therapeutics that showed evidence of efficacy to increase level of consciousness and functional communication in some Minimally Conscious State (MCS) patients, and in some Vegetative State (VS) patients. However the optimal intensity of electrical current stimulation remains unknown and transcranial Alternative Current Stimulation (tACS), with the ability to stimulate cortex at specific frequencies and to manipulate phase-synchrony between regions is a promising techniques to improve patients' consciousness.

In this study, the investigators will use prefrontal tDCS and theta tACS to improve patients consciousness level.

DETAILED DESCRIPTION:
This study is constituted of two independent sub-studies investigating two types of stimulation (tDCS and tACS) with the same cross-over design

Study design The study design is composed of two experimental sessions, one active stimulation and one sham comparator. Sessions will be randomized in a double-blind randomized crossover design (neither the participant nor the experimenter knows which session includes which stimulation type), with at least 2 days of interval between them.

In these sessions, the patients' state of consciousness participants will first be determined using the dedicated Coma Recovery Scale - Revised (Giacino, Neurology 2002) (CRS-R) scale before stimulation. Resting state brain activity EEG and cognitive auditory paradigm (local-global paradigm, Bekinschtein, PNAS 2009) will also be recorded before stimulation.

Twenty minutes stimulation will then be performed (see below). CRS-R, resting state EEG and local-global paradigm will be repeated after stimulation.

Outcome measures will be the same in the two studies. The primary outcome will be the change of CRS-R between before and after stimulation. Secondary outcomes will be the neurophysiological correlates of consciousness in resting state EEG and during the local global paradigm.

tACS stimulation During tACS sessions, 6 Hz stimulation (1000 μA) will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) using an 8-channels stimulator (Starstim NE, Neuroelectrics, Barcelona, Spain) with small round sponge electrodes (25 cm2 surface, maximal current density of 0.06 μA/cm2), controlled via Bluetooth. In the in-phase condition, the phase difference between the two stimulation sites will be 0° which will entrain synchronization between sites. In the sham condition, the stimulation will start with a current intensity of 1000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. Each stimulation session will take 20 minutes and the positions of stimulation electrodes and the duration of the stimulation will be kept identical for all conditions.

tDCS stimulation During tDCS session, 2000 μA stimulation will be applied over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) (Starstim NE, Neuroelectrics, Barcelona, Spain) with small round sponge electrodes (25 cm2 surface, maximal current density of 0.06 μA/cm2), controlled via Bluetooth. In the sham condition, the stimulation will start with a current intensity of 2000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. Each stimulation session will take 20 minutes and the positions of stimulation electrodes and the duration of the stimulation will be kept identical for all conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Non communicative patients with disorder of consciousness diagnosed by CRS-R (VS, MCS, exitMCS)
* Patients with stable clinical examination (even in intensive care)
* Brain injury confirmed by cerebral imaging (MRI or TDM)
* French social security affiliation
* Signed and informed consent by the patient or by a legal representant

Exclusion Criteria:

* Status epilepticus or uncontrolled epilepsy
* Severely neurodegenerative illnesses (Alzheimer disease, Lewy Body Dementia)
* Electrical stimulation contraindication (metallic intra-cranial implants, pacemaker or implantable cardioverter-defibrillator, cranial prosthesis)
* Pregnant, parturient or breastfeeding women- Patients underage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
State of consciousness | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change of the Coma Recovery Scale-Revised scores (CRS-R, Giacino et al. Neurology 2002 and Kalmar et al., Neuropsychol Rehabil 2005) between before and after stimulation (CRS-R post stimulation - CRS-R before stimulation). The CRS-R score is a qualitative and quantitative scales ranking predefined behaviors elicited by the patients in the following six subscales, auditory function, visual function, motor function, verbal and oromotor function, communication and wakefulness, the sum of which give a total score ranging from 0 to 23. Higher values of the scale mean a better state of consciousness. This change in state of consciousness will be compared between active stimulation and sham stimulation

SECONDARY OUTCOMES:
Evoked response potential during local-global paradigm | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change of the ERPS recorded during the "local global" auditory paradigm (Bekinschtein et al., PNAS 2009)
Resting state EEG | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change from baseline of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain et al. 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo D Sitt, MD, PhD, Principal Investigator — CR-ICM U 975 /UMRS INSERM 1127; Lionel Naccache, MD, PhD, Principal Investigator — CR-ICM U 975 /UMRS INSERM 1127; Bertrand Hermann, MD, Principal Investigator — CR-ICM U 975 /UMRS INSERM 1127
Locations (1):
- Institut du Cerveau et de la Moelle - CR-ICM U 975 / UMRS INSERM 1127, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Kalmar K, Giacino JT. The JFK Coma Recovery Scale--Revised. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):454-60. doi: 10.1080/09602010443000425. PMID 16350986